CLINICAL TRIAL: NCT01109511
Title: A Comparison of Oxycodone/Naloxone and Oxycodone After Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Mundipharma AB (Industry)
Responsible Party: Principal Investigator, Johan C Ræder, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: targiniqoxycodulleval
Record Dates: First submitted 2010-04-15; First posted 2010-04-23 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain; Opioid Induced Constipation
MeSH Terms: conditions — Pain, Postoperative; Opioid-Induced Constipation | interventions — Naloxone; Oxycodone

ARMS (2):
- oxycodone+naloxone (Active Comparator)
  Interventions: Drug: naloxone; Drug: oxycodone
- Control (Active Comparator): Oxycodone alone without naloxone
  Interventions: Drug: oxycodone

INTERVENTIONS:
Drug: naloxone
  Arms: oxycodone+naloxone
Drug: oxycodone

SUMMARY:
Objectives:

Primary objective:

* To demonstrate that the treatment with OXN PR tablets up to 72 hrs after surgery is superior to the treatment with OxyPR with regards to constipation in subjects with postoperative pain after laparoscopic hysterectomy based on interviews 24h, 72 h and 1 week postoperatively.

The secondary objectives:

* Analgesic effect (including registration during the first 24 hrs)
* To asses the frequency of pain rescue mediation use (in the double-blind phase, 0-72 hrs)
* Frequency of nausea and vomiting
* Frequency of other adverse events
* Appetite
* Mobilization

The exploratory objectives:

* Overall patient satisfaction at 24, 72 hrs and 1 week

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 -70 years
2. Elective, non-malignant laparoscopic gynecological surgery in general anesthesia : hysterectomy/ myomectomy, ASA 1, 2 and 3
3. Subjects willing and able to participate the study and have provided informed consent form -

Exclusion Criteria:

1. Previous recent or regular opioid use (WHO step I pain treatment allowed)
2. Any situation where opioids are contraindicated.
3. Any history of moderate to severe hepatic impairment.
4. Any history of severe respiratory depression with hypoxia and/or hypercapnia
5. Any history of severe chronic obstructive pulmonary disease, cor pulmonal, acute severe bronchial asthma
6. Subjects with evidence of non-opioid induced paralytic ileus
7. Subjects with evidence of severely impaired pulmonary function, myxoedema, hypothyroidism
8. Subjects with evidence of Addison's disease (adrenal cortical insufficiency), toxic psychosis,cholelithiasis, prostate hypertrophy, alcoholism, delirium, pancreatitis, hypotension, hypertension, pre-existing cardiovascular diseases, head injury (due to the risk of increased intracranial pressure), epileptic disorder or predisposition to convulsions, or patients taking MAO inhibitors.
9. Any history of hypersensitivity to Oxycodone / Naloxone or to any of the excipients.
10. Active alcohol or drug abuse and/or history of opioid abuse.
11. Subjects with evidence of clinically unstable disease, as determined by medical history, clinical laboratory tests, ECG results, and physical examination that, in the Investigator's opinion, preclude entry into the study.
12. Subjects who have received an investigational medicinal product within 30 days of study entry (defined as the start of the Screening Period).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-07-30 (Actual)

PRIMARY OUTCOMES:
Constipation in subjects with postoperative pain | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology, Oslo University Hospital, Ullevaal, Oslo, Norway